CLINICAL TRIAL: NCT02552615
Title: Investigation of the Effects of Spinal Stabilization and Body Awareness Exercises on Subjective Vertical Perception, Curve Magnitude, Body Symmetry and Quality of Life in Adolescent Idiopathic Scoliosis
Brief Title: Effectiveness of Exercises in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gözde Gür (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Gözde Gür, research assistant, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Go 14/19
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: scoliosis, verticality perception, body symmetry
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- body awareness therapy (BAT) (Experimental): Each session started with short warm-up, continued with specific exercises. Following each session, verbal reflexions was taken for 10 minutes. Exercises fulfilled in lying, sitting, standing and walking positions. Additionally program included vocal-breathing exercises and massage. Patients received 20 sessions for one hour at clinic for ten-week treatment period.
  Interventions: Other: body awareness therapy
- Traditional exercises (Active Comparator): Program included traditional exercises intended for strengthening back, abdominal, pelvis and shoulder girdle muscles and muscles in convex side of the curve, stretching exercises especially for the concave side of the curve, flexibility exercises for spine, postural training and breathing exercises. Patients received 20 sessions for one hour at clinic for ten-week treatment period.
  Interventions: Other: traditional exercises
- core stabilization exercises (Experimental): Exercises started to progress from static to dynamic positions in which muscle activation incorporate into functional tasks including trunk and extremity movements. Local, global muscle stability training, global muscle mobility training and strengthening training of these core structure was carried out progressively advancing more difficult. Patients received 20 sessions for one hour at clinic for ten-week treatment period.
  Interventions: Other: core stabilization exercises

INTERVENTIONS:
Other: body awareness therapy
  Arms: body awareness therapy (BAT)
Other: core stabilization exercises
  Arms: core stabilization exercises
Other: traditional exercises
  Arms: Traditional exercises

SUMMARY:
The aim of this study was to compare the effects of spinal stabilization and body awareness in addition to brace wearing versus classical exercises on subjective verticality perception, trunk symmetry and quality of life in AIS. Study included 30 AIS patients between the ages of 14.40±201 years (stabilization group), 14.2±2 years (Body awareness) and 13.60±1.65 (classical). Cobb angles, rotation, subjective visual (SVV), postural (SPV) and haptic (SHV) and deformity perception, quality of life were assessed at baseline and after 10th week of treatment. Cobb angle decreased in stabilization and awareness groups. Rotation decreased in three groups. SVV improved in all groups. SPV and SHV, body asymmetry and cosmetic deformity improved in stabilization and awareness groups. Only function improved with stabilization treatment. Stabilization and body awareness exercises created positive changes in AIS.

DETAILED DESCRIPTION:
In patients with idiopathic scoliosis (IS), in addition to curve progression there are many problems including altered posture, gait deviations, muscular imbalance, functional limitations, back pain, negative physico-social, body image effects, and in severe cases pulmonary symptoms commonly occur. To cope with these complications and more, conservative treatment of adolescent idiopathic scoliosis (AIS) involves a variety of bracing methods and exercises.

Spinal bracing is an important treatment option to prevent curve progression in moderate curves (between 20-40) and severe curves in AIS. Bracing success rate is reported 80% in the long term but the level of evidence is still low.

In literature, exercises are recommended to reduce progression, to improve spine and thoracic cage flexibility, muscle elasticity and strength, to correct postural behavior, and neuro-motor control, spine stability. In general, traditional exercises (TE) including stretching, strengthening exercises for spinal musculature, postural training, respiratory exercises have been used for many years for IS. Besides traditional exercises, there are several exercise concepts including SEAS, Schroth, Dobomed, Side Shift methods... etc. Effectiveness of exercise is still in debate and there is need for further studies, which investigate the role of specific exercises for scoliosis in conservative treatment.

In scoliosis, muscle imbalances, the deficiency of muscle ability to stabilize posture, the loss in balance of pelvis-spine relation due to lateral tilt of the body and postural control impairment resulting from these problems are defined. In addition, the tree dimensional scoliotic deformity cause sensory disturbances, standing instability and gait modifications. Core stabilization exercises (CSE) are described as therapy technique that improve neuromuscular control, strength of trunk stabilization muscles, endurance of postural muscles, trunk mobilization muscles around spine, balance between pelvis and spine in order to maintain functional stability and postural control.

It was indicated in the literature that patients with AIS exhibit disturbances of vertical perception. Postural vertical line is important for a person to perceive body orientation in space and thereby to provide and maintain upright posture and gait. Body Awareness Therapy (BAT) is a mind-body approach, which aims to improve body awareness, body posture, quality of movements, balance, postural control integrating with slow movement co-ordination and breathing exercises. BAT programs also contain stretching exercises, relaxing exercises and gait training. Patients are instructed to concentrate body vertical line and all movements are thought to initiate from body center. BAT have been studied in many medical conditions including back pain, anxiety, fibromyalgia, eating disorders, heart diseases, falls in elderly.

However, there are limited studies determining CSE effects on patients with scoliosis: one have reported improvement in Cobb's angle and pain and the other in sitting balance with lumbar stabilization exercises. There was no research examining the effects of BAT in scoliosis. However for the reasons mentioned above, we hypothesized that CSE and BAT therapies can have positive effects on postural re-alignment and trunk deformity in patients with AIS. The aim of this study was to investigate the effects of core stabilization and body awareness exercises versus traditional exercises in addition to brace wearing on vertical perception, trunk asymmetry, cosmetic deformity and health related quality of life in patients with AIS.

The aim of this study was to compare the effects of spinal stabilization and body awareness exercises in addition to brace wearing versus traditional exercises on subjective verticality perception, trunk symmetry, cosmetic deformity and health related quality of life in Adolescent idiopathic scoliosis (AIS). This study included 30 AIS patients between the ages of 14,40 ± 2,01 years (stabilization group), 14,2 ± 2 years (Body awareness group) ve 13,60 ± 1,65 (classical group). Following recording demographic data, bone maturation level according to Riser, curve types according to King, spinal region, which includes curve, were recorded. Cobb angles by antero-posterior X-ray, rotation degrees with scoliometer in Adam's forward bend test, subjective visual (SVV), postural (SPV) and haptic (SHV) verticality perception with laser stick system, cosmetic deformity perception for patient, family and physiotherapist according with Walter Reed Visual Assessment Scale (WRVAS), trunk asymmetries with Posterior Trunk Asymmetry Index (POTSI) and health related quality of life with SRS-22 were assessed at baseline and after 10th week of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed with idiopathic scoliosis
* ages between 10 and 16 who were prescribed a brace

Exclusion Criteria:

* Patients who did not accept to participate in the study or wear a spinal brace
* congenital curve
* neuromuscular, rheumatologic, renal, cardiovascular, pulmonary or vestibular diseases, tumors,
* previous surgical correction or conservative therapy

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cobb angle | 10 weeks
  Cobb's angles were measured on standard standing anterior-posterior spine radiograph and recorded as degrees. Cobb angle is considered the gold standard to evaluate the curve magnitude

SECONDARY OUTCOMES:
Posterior Trunk Asymmetry Index (POTSI) | 10 weeks
  POTSI is a surface topography method, which scores body shape and asymmetry objectively. The measurements of patient's back were taken for the calculation of the score POTSI is composed of six index including frontal asymmetry index (FAI), height differences index (HDI) for shoulder, axilla and trunk regions. Total score is a sum of these six indexes.
axial trunk rotation | 10 weeks
  Axial trunk rotations (ATR) were assessed with scoliometer in Adam's forward bend test
Walter Reed Visual Assessment Scale (WRVAS) | 10 weeks
  WRVAS was used to assess cosmetic deformity. The domains of WRVAS are body curve, rib prominence, flank prominence, head rib pelvis, head pelvis, shoulder level and scapular rotation. Each domain generates a score from 1 (best deformity) to 5 (worst deformity). Total score is an average of these 7 domains
SRS-22 Questionnaire | 10 weeks
  It assess quality of life in scoliosis. This instrument consists of six domains including function, pain, self-image, mental health, satisfaction/dissatisfaction which are scored from 1 (best answer) to 5 (worst answer) each question
vertical perception | 10 weeks
  All visual (SVV), postural (SPV) and haptic (SHV) subjective vertical perception tests were performed using manually controlled laser liner device by the therapist in a darkened, silent and empty room. The therapist put laser line as deviated from vertical, then turned it to vertical slowly and asked patient to find true earth vertical. Subjects were instructed to tell "stop" when they thought it is correct angle for them. Assessment were repeated for horizontal line and at the angles of 30°, 45°, 60° left and 30°, 45°, 60° right (according to the ground). This test expressed SVV assessment. For SPV patient predict angle with his/her hand position. For SHV, patients predict angle by holding a wooden stick with their hands.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Gur, PhD, Principal Investigator — research assistant and physiotherapist
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

REFERENCES:
- [Background] Romano M, Minozzi S, Zaina F, Saltikov JB, Chockalingam N, Kotwicki T, Hennes AM, Negrini S. Exercises for adolescent idiopathic scoliosis: a Cochrane systematic review. Spine (Phila Pa 1976). 2013 Jun 15;38(14):E883-93. doi: 10.1097/BRS.0b013e31829459f8. PMID 23558442
- [Background] Yang JH, Suh SW, Sung PS, Park WH. Asymmetrical gait in adolescents with idiopathic scoliosis. Eur Spine J. 2013 Nov;22(11):2407-13. doi: 10.1007/s00586-013-2845-y. Epub 2013 Jun 4. PMID 23732766
- [Background] Shneerson JM, Madgwick R. The effect of physical training on exercise ability in adolescent idiopathic scoliosis. Acta Orthop Scand. 1979 Jun;50(3):303-6. doi: 10.3109/17453677908989771. PMID 474101
- [Background] Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Effects of bracing in adolescents with idiopathic scoliosis. N Engl J Med. 2013 Oct 17;369(16):1512-21. doi: 10.1056/NEJMoa1307337. Epub 2013 Sep 19. PMID 24047455
- [Background] Maruyama T, Grivas TB, Kaspiris A. Effectiveness and outcomes of brace treatment: a systematic review. Physiother Theory Pract. 2011 Jan;27(1):26-42. doi: 10.3109/09593985.2010.503989. PMID 21198404
- [Background] Negrini S, Minozzi S, Bettany-Saltikov J, Chockalingam N, Grivas TB, Kotwicki T, Maruyama T, Romano M, Zaina F. Braces for idiopathic scoliosis in adolescents. Cochrane Database Syst Rev. 2015 Jun 18;2015(6):CD006850. doi: 10.1002/14651858.CD006850.pub3. PMID 26086959
- [Background] Negrini S, Fusco C, Minozzi S, Atanasio S, Zaina F, Romano M. Exercises reduce the progression rate of adolescent idiopathic scoliosis: results of a comprehensive systematic review of the literature. Disabil Rehabil. 2008;30(10):772-85. doi: 10.1080/09638280801889568. PMID 18432435
- [Background] Nault ML, Allard P, Hinse S, Le Blanc R, Caron O, Labelle H, Sadeghi H. Relations between standing stability and body posture parameters in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1911-7. doi: 10.1097/00007632-200209010-00018. PMID 12221357
- [Background] Muthukrishnan R, Shenoy SD, Jaspal SS, Nellikunja S, Fernandes S. The differential effects of core stabilization exercise regime and conventional physiotherapy regime on postural control parameters during perturbation in patients with movement and control impairment chronic low back pain. Sports Med Arthrosc Rehabil Ther Technol. 2010 May 31;2:13. doi: 10.1186/1758-2555-2-13. PMID 20515453
- [Background] Cakrt O, Slaby K, Viktorinova L, Kolar P, Jerabek J. Subjective visual vertical in patients with idiopatic scoliosis. J Vestib Res. 2011;21(3):161-5. doi: 10.3233/VES-2011-0414. PMID 21558641
- [Background] Alves de Araujo ME, Bezerra da Silva E, Bragade Mello D, Cader SA, Shiguemi Inoue Salgado A, Dantas EH. The effectiveness of the Pilates method: reducing the degree of non-structural scoliosis, and improving flexibility and pain in female college students. J Bodyw Mov Ther. 2012 Apr;16(2):191-8. doi: 10.1016/j.jbmt.2011.04.002. Epub 2012 Jan 5. PMID 22464116
- [Background] Gur G, Dilek B, Ayhan C, Simsek E, Aras O, Aksoy S, Yakut Y. Effect of a spinal brace on postural control in different sensory conditions in adolescent idiopathic scoliosis: a preliminary analysis. Gait Posture. 2015 Jan;41(1):93-9. doi: 10.1016/j.gaitpost.2014.09.001. Epub 2014 Sep 16. PMID 25262334
- [Background] Coelho DM, Bonagamba GH, Oliveira AS. Scoliometer measurements of patients with idiopathic scoliosis. Braz J Phys Ther. 2013 Mar-Apr;17(2):179-84. doi: 10.1590/S1413-35552012005000081. PMID 23778766
- [Background] Sanders JO, Polly DW Jr, Cats-Baril W, Jones J, Lenke LG, O'Brien MF, Stephens Richards B, Sucato DJ; AIS Section of the Spinal Deformity Study Group. Analysis of patient and parent assessment of deformity in idiopathic scoliosis using the Walter Reed Visual Assessment Scale. Spine (Phila Pa 1976). 2003 Sep 15;28(18):2158-63. doi: 10.1097/01.BRS.0000084629.97042.0B. PMID 14501929
- [Background] Monticone M, Ambrosini E, Cazzaniga D, Rocca B, Ferrante S. Active self-correction and task-oriented exercises reduce spinal deformity and improve quality of life in subjects with mild adolescent idiopathic scoliosis. Results of a randomised controlled trial. Eur Spine J. 2014 Jun;23(6):1204-14. doi: 10.1007/s00586-014-3241-y. Epub 2014 Feb 28. PMID 24682356
- [Background] Rumsey N, Harcourt D. Body image and disfigurement: issues and interventions. Body Image. 2004 Jan;1(1):83-97. doi: 10.1016/S1740-1445(03)00005-6. PMID 18089143
- [Background] Mehling WE, Wrubel J, Daubenmier JJ, Price CJ, Kerr CE, Silow T, Gopisetty V, Stewart AL. Body Awareness: a phenomenological inquiry into the common ground of mind-body therapies. Philos Ethics Humanit Med. 2011 Apr 7;6:6. doi: 10.1186/1747-5341-6-6. PMID 21473781
- [Background] Bisdorff AR, Wolsley CJ, Anastasopoulos D, Bronstein AM, Gresty MA. The perception of body verticality (subjective postural vertical) in peripheral and central vestibular disorders. Brain. 1996 Oct;119 ( Pt 5):1523-34. doi: 10.1093/brain/119.5.1523. PMID 8931577
- [Background] Seferiadis A, Ohlin P, Billhult A, Gunnarsson R. Basic body awareness therapy or exercise therapy for the treatment of chronic whiplash associated disorders: a randomized comparative clinical trial. Disabil Rehabil. 2016;38(5):442-51. doi: 10.3109/09638288.2015.1044036. Epub 2015 May 8. PMID 25955823
- [Background] Danielsson L, Papoulias I, Petersson EL, Carlsson J, Waern M. Exercise or basic body awareness therapy as add-on treatment for major depression: a controlled study. J Affect Disord. 2014 Oct;168:98-106. doi: 10.1016/j.jad.2014.06.049. Epub 2014 Jul 5. PMID 25043321